CLINICAL TRIAL: NCT03799783
Title: The Use of Dexmedetomidine for Procedural Sedation During EEG in Children Affected by Behavioural Disorders
Brief Title: The Use of Dexmedetomidine for EEG Sedation in Children With Behavioural Disorders
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Azienda Ospedaliera di Padova (Other)
Responsible Party: Principal Investigator, angela amigoni, Principal Investigator, Azienda Ospedaliera di Padova
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4422/AO/18
Record Dates: First submitted 2019-01-03; First posted 2019-01-10 (Actual); Results first posted 2021-01-15 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Procedural Sedation; Behavior Disorders
Keywords: dexmedetomidine; sedation
MeSH Terms: conditions — Mental Disorders | interventions — Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: Drug administration by a loading dose followed by continuous infusion during a procedure
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dexmedetomidine (Experimental): 2 mcg/Kg iv dexmedetomidine (this dose may be repeated up to 2 times) followed by 1-2 mcg/Kg/hour iv continuous infusion
  Interventions: Drug: dexmedetomidine

INTERVENTIONS:
Drug: dexmedetomidine — To administer dexmedetomidine IV 2 μg/kg in 10 minutes (loading dose) followed by continuous infusion at a rate of 1 μg/kg/h until procedure was complete
  Other Names: dexdor

SUMMARY:
Children's compliance during diagnostic or therapeutic procedures is a challenge, often requiring the use of sedative and/or analgesic drugs.

Electroencephalogram (EEG) needs stillness for a medium-long period but, at the same time, the use of any drug for sedation may affect the exam through an interference with EEG waves. Dexmedetomidine is a selective ∝2-adrenergic agonist with sedative and anxiolytic properties, with a long effect and which does not alter EEG pattern.

The aim of this interventional study is to evaluate the effectiveness, safety and feasibility of dexmedetomidine for sedation during EEG in children who are not cooperative.

Children affected by behavioral disorders and requiring sedation to perform EEG were considered. The protocol establishes to administer IV dexmedetomidine (loading dose and continued infusion) to reach a targeted level of sedation (Pediatric Sedation State Scale = 2). Vital signs (SatO2, RR, EtCO2, HR, BP) and level of sedation are recorded before, during and after procedure until the offset.

DETAILED DESCRIPTION:
Compliance during diagnostic or therapeutic procedures is a very frequent challenge in children. Procedural sedation and analgesia represents an effective answer to this problem. Electroencephalogram (EEG) is a procedure which needs stillness for a medium-long period. Whereas the majority of children carry out this procedure without sedation, patients with behavioral problems, who frequently need to rule out the presence of seizures as associated symptoms or different disease, often show an insufficient compliance. Sedative drugs usually interfere with EEG cerebral waves pattern, so they can not be used. Dexmedetomidine is a selective ∝2-adrenergic agonist with prevalent sedative and anxiolytic properties, with a long effect and which does not alter EEG pattern.

The aim of this interventional study is to evaluate effectiveness, safety and feasibility of dexmedetomidine for sedation during EEG in children who are not cooperative.

Children referred to the Pediatric Neurology Department of the Pediatric Hospital of Padova and required sedation to perform EEG were considered in the study.

The protocol establishes to administer dexmedetomidine IV 2 μg/kg in 10 minutes (loading dose) followed by continuous infusion at a rate of 1 μg/kg/h until procedure was complete. The loading dose can be repeated up to two times, if needed, to achieve the targeted level of Pediatric Sedation State Scale (PSSS) of 2 (quiet, asleep or awake, not moving during procedure, and no frown or brow furrow indicating pain or anxiety, no verbalization of any complaint). Vital signs (SatO2, RR, EtCO2, HR, BP) and level of sedation are recorded before, during and after procedure until the complete awake of the patient. The quality of the EEG pattern was also evaluated. Occurrence and type of adverse events are registered during this period. Finally, the caregivers' opinion about the quality of the sedation and the presence of any sleep disturbance at home during the next 12 hours after the procedure were considered.

ELIGIBILITY:
Inclusion Criteria:

* children affected by behavior disorders who underwent EEG procedure with sedation
* written informed consent

Exclusion Criteria:

* ASA > 2
* hypersensitivity of active substance
* therapy with beta blockers or digoxin, arrhythmia

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 19 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: angela amigoni, MD, Principal Investigator — azienda Ospedaliera di Padova-Pediatric Intensive Care Unit
Locations (1):
- Pediatric Intensive Care Unit - Department of Woman's and Child's Health - Azienda Ospedaliera di Padova, Padua, PD, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mason KP, O'Mahony E, Zurakowski D, Libenson MH. Effects of dexmedetomidine sedation on the EEG in children. Paediatr Anaesth. 2009 Dec;19(12):1175-83. doi: 10.1111/j.1460-9592.2009.03160.x. PMID 20017865
- [Result] Cravero JP, Askins N, Sriswasdi P, Tsze DS, Zurakowski D, Sinnott S. Validation of the Pediatric Sedation State Scale. Pediatrics. 2017 May;139(5):e20162897. doi: 10.1542/peds.2016-2897. PMID 28557732
- [Result] National Clinical Guideline Centre (UK). Sedation in Children and Young People: Sedation for Diagnostic and Therapeutic Procedures in Children and Young People [Internet]. London: Royal College of Physicians (UK); 2010 Dec. Available from http://www.ncbi.nlm.nih.gov/books/NBK82237/ PMID 22536619
- [Result] Cote CJ, Wilson S; AMERICAN ACADEMY OF PEDIATRICS; AMERICAN ACADEMY OF PEDIATRIC DENTISTRY. Guidelines for Monitoring and Management of Pediatric Patients Before, During, and After Sedation for Diagnostic and Therapeutic Procedures: Update 2016. Pediatrics. 2016 Jul;138(1):e20161212. doi: 10.1542/peds.2016-1212. PMID 27354454
- [Result] Sulton C, McCracken C, Simon HK, Hebbar K, Reynolds J, Cravero J, Mallory M, Kamat P. Pediatric Procedural Sedation Using Dexmedetomidine: A Report From the Pediatric Sedation Research Consortium. Hosp Pediatr. 2016 Sep;6(9):536-44. doi: 10.1542/hpeds.2015-0280. Epub 2016 Aug 11. PMID 27516413
- [Result] Keidan I, Ben-Menachem E, Tzadok M, Ben-Zeev B, Berkenstadt H. Electroencephalography for children with autistic spectrum disorder: a sedation protocol. Paediatr Anaesth. 2015 Feb;25(2):200-5. doi: 10.1111/pan.12510. Epub 2014 Aug 22. PMID 25145661
- [Result] Lubisch N, Roskos R, Berkenbosch JW. Dexmedetomidine for procedural sedation in children with autism and other behavior disorders. Pediatr Neurol. 2009 Aug;41(2):88-94. doi: 10.1016/j.pediatrneurol.2009.02.006. PMID 19589455
- [Result] Zub D, Berkenbosch JW, Tobias JD. Preliminary experience with oral dexmedetomidine for procedural and anesthetic premedication. Paediatr Anaesth. 2005 Nov;15(11):932-8. doi: 10.1111/j.1460-9592.2005.01623.x. PMID 16238552

RESULTS

PARTICIPANT FLOW:
Groups:
- Dexmedetomidine: 2 mcg/Kg iv dexmedetomidine (this dose may be repeated up to 2 times) followed by 1-2 mcg/Kg/hour iv continuous infusion
  dexmedetomidine: To administrater dexmedetomidine IV 2 μg/kg in 10 minutes (loading dose) followed by continuous infusion at a rate of 1 μg/kg/h until procedure was complete
Period: Overall Study
Arm/Group | Dexmedetomidine
Started | 19
Completed | 19
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Dexmedetomidine
Number analyzed (Participants) | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.3 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients That Reach a Score Equal or Lower Than 2 Ten Minutes After the Infusion of Dexmedetomidine (Assessed With the PSSS Pediatric Sedation State Scale)
Description: the PSSS is a validated scale for assessing the level of procedural sedation. It is a 6 items scale , from 0 to 5, where 5 is an alert patient and 0 is a deep sedation with abnormal vital signs. We evaluate patients 10 minutes after the infusion of dexmedetomidine.
Time Frame: 10 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Dexmedetomidine
Number analyzed (Participants) | 19
Participants | 13

2. Secondary Outcome: Number of Patients With Adverse Events
Description: any adverse event potentially related with DEX-administration
Time Frame: during and immediately after DEX infusion, up to 150 minutes after DEX infusion (time to first awakening)
Measure: Count of Participants; unit: Participants
Arm/Group | Dexmedetomidine
Number analyzed (Participants) | 19
Participants | 10

ADVERSE EVENTS:
Time Frame: 90 minutes
Description: Other (not including serious) adverse events
Arm/Group | Dexmedetomidine
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 10/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dexmedetomidine (N=19)
hypotension (Cardiac disorders) | 6 (6) — spontaneously resolved
bradycardia (Cardiac disorders) | 4 (4) — spontaneously resolved

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-20): https://cdn.clinicaltrials.gov/large-docs/83/NCT03799783/Prot_SAP_000.pdf